CLINICAL TRIAL: NCT06747130
Title: Efficacy of Montelukast in Preventing Transaminase Elevation in Adult Dengue Patients: a Randomized, Double-blind, Placebo Controlled, Superiority Trial
Brief Title: Efficacy of Montelukast in Preventing Transaminase Elevation in Adult Dengue Patients
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Phramongkutklao College of Medicine and Hospital (Other)
Responsible Party: Principal Investigator, Vasin Vasikasin, Assistant Professor, Consultant in Infectious Disease, Phramongkutklao College of Medicine and Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R165h/67
Record Dates: First submitted 2024-12-18; First posted 2024-12-24 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Dengue; Montelukast; Transaminases
MeSH Terms: conditions — Dengue | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Montelukast (Experimental): a 10 mg tablet will be given orally immediately and every day thereafter for 10 days or until recovery, defined as the discontinuation of the follow up appointment by the attending physicians, whichever is shorter
  Interventions: Drug: Montelukast
- Placebo (Placebo Comparator): a 10 mg tablet will be given orally immediately and every day thereafter for 10 days or until recovery, defined as the discontinuation of the follow up appointment by the attending physicians, whichever is shorter
  Interventions: Drug: Montelukast Placebo

INTERVENTIONS:
Drug: Montelukast — A 10-mg tablet will be given orally immediately and every day thereafter for 10 days or until recovery, defined as the discontinuation of the follow up appointment by the attending physicians, whichever is shorter
  Arms: Montelukast
Drug: Montelukast Placebo — A 10-mg tablet will be given orally immediately and every day thereafter for 10 days or until recovery, defined as the discontinuation of the follow up appointment by the attending physicians, whichever is shorter
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if drug montelukast works to treat dengue in adults. It will also learn about the safety of drug montelukast . The main questions it aims to answer are:

Does drug montelukast lower the incidence of liver enzyme elevations in participants ? What medical problems do participants have when taking drug montelukast ?

DETAILED DESCRIPTION:
Dengue remains a significant and growing public health issue in many tropical countries, with almost 4 billion people estimated to be at risk worldwide and an annual incidence of approximately 400 million infections. In 2019 alone, 5.2 million cases of dengue were reported globally.

In addition to its acute clinical manifestations, dengue is a leading cause of liver failure in tropical regions. Elevated concentrations of transaminases have been strongly correlated with disease severity. Severe acute hepatitis in dengue patients is associated with prolonged hospital stays, increased mortality, bleeding complications, and renal failure. While transaminase elevations are commonly linked to shock and subsequent ischemic hepatitis, studies indicate that these elevations often precede the onset of shock by several days. Notably, elevated transaminase levels during the febrile stage have been predictive of subsequent shock, underscoring their potential role as an early marker of disease progression.

Leukotrienes play a pivotal role in the pathophysiology of dengue by promoting plasma leakage and leukocyte adhesion within postcapillary venules. In dengue patients, leukotriene levels are markedly elevated-up to 35-38 times baseline levels-during the febrile and defervescence stages, returning to normal during the convalescent phase. Animal model studies have demonstrated that leukotriene blockade significantly reduces plasma leakage, suggesting its potential as a therapeutic target.

Currently, the management of dengue is limited to symptomatic treatment and intravenous fluid replacement, with no specific interventions proven to prevent complications. Preclinical studies have identified nafamostat, a tryptase inhibitor, and montelukast, a leukotriene receptor antagonist, as promising agents for reducing plasma leakage. An open-label clinical study in 2018 reported a 22% absolute risk reduction in dengue shock syndrome among patients treated with montelukast compared to standard care. However, a subsequent randomized controlled trial in 2024 failed to demonstrate efficacy of montelukast in preventing plasma leakage or warning signs of severe dengue. This discrepancy may reflect either the ineffectiveness of montelukast or the low incidence of warning signs in the trial population. Interestingly, secondary analyses revealed that participants in the montelukast group had a lower incidence of transaminase elevations compared to those receiving placebo, suggesting a potential hepatoprotective effect.

This study aims to evaluate the efficacy of montelukast in reducing the incidence of transaminase elevations in adult patients with dengue.

ELIGIBILITY:
Inclusion Criteria:

* Patient age >18 years
* Dengue infection diagnosed by NS1 antigen, or polymerase chain reaction
* Admitted to the hospital
* Written informed consent from patient or attending relative able to and willing to give informed consent

Exclusion Criteria:

* Other possible cause of fever other than dengue infection
* Pregnancy
* Unable to take medication
* Aminotransferase level above 150 U/l
* Allergy to paracetamol or tramadol
* Paracetamol indicated for condition other than dengue infection
* Critically ill patient who need ICU or invasive ventilation support
* History of cirrhosis
* Unable to communicate
* Other indication of montelukast
* History of psychiatric illness

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2025-01-31 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Serum transaminase levels on the recovery day | From enrollment to the end of treatment at 10 days
  Serum alanine transaminase and aspartate transaminase level will be measured at admission, and on every morning afterwards until the subject is discharged. The proportion of subjects with abnormal serum transaminase levels will be compared. The recovery day is defined as the day the participant was discharged from the hospital.

SECONDARY OUTCOMES:
Proportion of subjects with abnormal serum transaminase levels on the recovery day | From enrollment to the end of treatment at 10 days
  Serum alanine transaminase and aspartate transaminase level will be measured at admission, and on every morning afterwards until the subject is discharged. The proportion of subjects with abnormal serum transaminase levels will be compared.
Length of stay | From enrollment to the end of treatment at 10 days
  Duration from hospital admission to discharge will be compared.
Changes in serum transaminase levels | From enrollment to the end of treatment at 10 days
  The change in serum transaminase levels from baseline at admission will be compared.
Rate of dengue with warning signs | From enrollment to the end of treatment at 10 days
  Rate of a composite outcome including abdominal tenderness or pain, persistent vomiting, clinical fluid accumulation, mucosal bleeding, liver enlargement >2cm, increase in hematocrit concurrent with decrease in platelet count
Rate of severe dengue | From enrollment to the end of treatment at 10 days
  Rate of a composite outcome including shock, fluid accumulation with respiratory distress, severe bleeding leading to hypotension or decreased hematocrit, liver transaminase >1000, impaired consciousness, heart and other organ failure
Rate of dengue shock | From enrollment to the end of treatment at 10 days
  Rate of hypotension or the pulse pressure of ≤ 20 mm Hg
Hematocrit and platelet | From enrollment to the end of treatment at 10 days
  Hematocrit and platelet levels will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Worapong Nasomsong, MD, Study Director — Phramongkutklao College of Medicine and Hospital
Locations (1):
- Phramongkutklao Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided